CLINICAL TRIAL: NCT00877175
Title: Comparison of Conventional Instillation and Lower Conjunctival Fornix Packing in Mydriasis for Premature Infants
Brief Title: Comparison of Instillation and Packing in Mydriasis for Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: I50221; HE480729
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Preterm Infants
Keywords: preterm infants; mydriasis; pupil dilation
MeSH Terms: conditions — Mydriasis | interventions — Tropicamide; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lower conjunctival fornix packing arm. For the eyes receiving lower conjunctival fornix packing (study group), one small piece of the cotton wool soaked with one drop of 2.5% phenylephrine and one drop of 1% tropicamide was packed in the lower conjunctival fornix.
  Interventions: Drug: 1% tropicamide and 2.5% phenylephrine
- 2 (Active Comparator): Conventional instillation arm. For the eyes receiving the instillation (control group), 2.5% phenylephrine and 1% tropicamide were alternately instilled every 5 minutes for two doses each.
  Interventions: Drug: 1% tropicamide and 2.5% phenylephrine

INTERVENTIONS:
Drug: 1% tropicamide and 2.5% phenylephrine — For the eyes receiving lower conjunctival fornix packing (study group), one small piece of the cotton wool soaked with one drop of 2.5% phenylephrine and one drop of 1% tropicamide was packed in the lower conjunctival fornix. For the eyes receiving the instillation (control group), 2.5% phenylephrine and 1% tropicamide were alternately instilled every 5 minutes for two doses each.

SUMMARY:
The purpose of this study is to compare the mydriatic effect of 2.5% phenylephrine and 1% tropicamide by conventional instillation and lower conjunctival fornix packing in premature infants.

DETAILED DESCRIPTION:
Adequate pupil dilatation was needed for screening and treatment of retinopathy of prematurity (ROP) in premature infants.In general clinical practice, mydriatic drugs were instilled many times until the pupil reached the maximum size. However, poor mydriasis were found in many eyes despite maximum instillation was used. From the clinical observation, we found the packing of mydriatic drugs in lower conjunctival fornix was much more effective to dilate the pupil than instillation in some patients. The purpose of this study was to compare the mydriatic effect of 2.5% phenylephrine and 1% tropicamide by conventional instillation and lower conjunctival fornix packing in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* gestational age of less than 32 weeks and/or the birth weight of less than 1,500 grams
* stable clinical course

Exclusion Criteria:

* history of intraocular surgery or laser treatment
* previous eyedrop instillation that might affect the pupil size
* severe underlying disease or unstable clinical course that mydriatic drugs or the examination could aggravate their conditions

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the horizontal pupil diameter measured with a ruler in millimeters | 40 minutes after mydriatric drugs

CONTACTS AND LOCATIONS:
Overall Officials: Yosanan Yospaiboon, M.D., Principal Investigator — Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Thanathanee O, Ratanapakorn T, Morley MG, Yospaiboon Y. Lower conjunctival fornix packing for mydriasis in premature infants: a randomized trial. Clin Ophthalmol. 2012;6:253-6. doi: 10.2147/OPTH.S28714. Epub 2012 Feb 15. PMID 22368443